CLINICAL TRIAL: NCT06200272
Title: Effect of Whole-Wheat Bread Enriched With Carob Molasse Pose Flour and Germ On Healthy Volunteers' Glycemic Response and Antioxidant Capacity
Brief Title: Effect of Carob Molasse Pose Flour and Germ On Glycemic Response and Antioxidant Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toros University (Other)
Responsible Party: Principal Investigator, Eda Parlak, Asst. Prof., Toros University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: EDA-YL-EBRAR-TOROS-001
Record Dates: First submitted 2023-12-13; First posted 2024-01-10 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
Keywords: Carob molasses pulp; germ; bread; glycemic load; antioxidant capacity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test group with standard whole wheat breads (Germ and Carob Molasses Pulp added) (Experimental): Bread will be produced by adding germ (obtained after processing the wheat grain), which has a high antioxidant capacity and is rich in vitamins and dietary fiber, and carob pulp (Carob Molasses Pulp, CMP), which is not considered waste after the production of carob molasses, to the formulation of wheat bread, which has been widely consumed in recent years.
  Interventions: Combination Product: Germ and Carob Molasses Pulp added standard whole wheat breads
- Control group with standard whole wheat breads (No Intervention): control bread (whole wheat bread) made based on a standard recipe

INTERVENTIONS:
Combination Product: Germ and Carob Molasses Pulp added standard whole wheat breads — Test bread (bread with soluble pulp added, bread with added germ, and bread with soluble pulp + germ added) containing 50 g carbohydrate, samples taken from all four types of bread were collected for moisture, ash, fiber, protein, fat, digestible carbohydrate, and antioxidant capacity analysis will be performed. This experimental group consists of the group that will eat the test bread.
  Arms: Test group with standard whole wheat breads (Germ and Carob Molasses Pulp added)

SUMMARY:
Test with standard whole wheat bread (germ and CMP added); Its effect on glycemic response and antioxidant capacity in healthy adults will be examined. For this purpose, adult individuals; will be carried out with 20 volunteer individuals between the ages of 19-35 years, who do not have acute or chronic diseases and whose Body Mass Index (BMI) value is between 18.5-24.9 kg/m2. Exclusion criteria will include using prescription drugs and/or nutritional supplements, being pregnant or lactating, excessive alcohol consumption (>2 drinks/day)/smoking, being in the menstrual period for female individuals, and being allergic to the foods to be used in the study. Individuals participating in the study will come to the research center twice in total, one week apart, to consume the bread produced. After eating their usual dinner the night before the test, individuals will be able to fast for 10-12 hours and drink only water during this period. Basal/fasting blood samples will be taken from individuals who come to the research center following fasting. The bread will be consumed within 10 minutes and venous blood samples will be taken by the nurse in charge at 30, 60, 120, and 180 minutes. During these three hours, individuals will be ensured not to leave the research center or consume any other food. Blood Glucose, Total Antioxidant Level (TAS), and Total Oxidant Level (TOS) values will be checked in the blood samples.

Blood Glucose, Total Antioxidant Level (TAS), and Total Oxidant Level (TOS) values will be statistically evaluated in the blood samples of individuals who consume standard whole wheat bread and the test whole wheat bread developed by us. If the results are found to be statistically significant, consuming the bread produced will play an important role in preventing chronic diseases such as obesity, diabetes, and cardiovascular diseases.

On the other hand; by adding CMP and germ, which are not currently evaluated, to the bread formulation, this study not only contributes to the prevention of food waste and sustainability by using low-cost food industry by-products but also enables the development of a bread-type with high nutritional value in terms of antioxidant-rich active ingredients, vitamins and dietary fiber.

DETAILED DESCRIPTION:
Bread is a traditional staple food widely consumed all over the world. In our country, whose diet is based on grain, the flour used in bread making is subjected to the refining process; The bran and germ parts are largely lost, resulting in a decrease in the nutritional value of the bread and an increase in the glycemic index and load. Therefore, consuming high amounts of bread containing refined flour has been associated with an increase in chronic diseases such as obesity, diabetes, and cardiovascular diseases. To reduce or eliminate this effect; In recent years, different nutritional enrichment studies aimed at reducing the health consequences mentioned above by improving the nutritional content of daily consumed bread have increasingly continued. In this study; Bread will be produced by adding germ (obtained after processing the wheat grain), which has a high antioxidant capacity and is rich in vitamins and dietary fiber, and carob pulp (Carob Molasses Pulp, CMP), which is not considered as waste after the production of carob molasses, to the formulation of whole wheat bread, which has been widely consumed in recent years. . The most suitable formulation will be determined by determining the chemical (moisture, ash, protein, fat, total and resistant starch, and antioxidant capacity) and sensory properties (appearance, crust color, taste, smell, chewiness, etc.) of the bread produced in this way.

ELIGIBILITY:
Inclusion Criteria:

* no acute or chronic disease
* no prescription drugs and/or nutritional supplements
* no pregnant or lactating
* no alcohol or excessive alcohol consumption (<2 drinks/day)
* no smoking,
* BMI value between 18.5-24.9 kg/m2
* no in the menstrual period for female individuals
* no gluten enteropathy
* no insulin resistance as a result of endocrinological examination and biochemical tests
* no allergic reaction to carob
* signed the Informed Volunteer Consent Form
* aged between 19 and 35 years.

Exclusion Criteria:

* having an acute or chronic disease
* using prescription drugs and/or nutritional supplements
* being in pregnancy and lactation
* consuming excessive alcohol (>2 drinks/day)
* smoking
* BMI value under 18.5 or above 24.9. kg/m2
* being in the menstrual period for female individuals
* having gluten enteropathy
* having insulin resistance as a result of endocrinological examination and biochemical tests
* having an allergic reaction to carob
* not signed the Informed Volunteer Form,
* aged under 19 years or above 35 years of age

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Whole wheat bread and blood glucose level at 0th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood glucose measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood glucose level at 0th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood glucose measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood TAS level at 0th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TAS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood TAS level at 0th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TAS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood TOS level at 0th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood TOS level at 0th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood glucose level at 30th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood glucose level at 30th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood TAS level at 30th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood TAS level at 30th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood TOS level at 30th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood TOS level at 30th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood glucose level at 60th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood glucose level at 60th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood TAS level at 60th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood TAS level at 60th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood TOS level at 60th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood TOS level at 60th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood glucose level at 120th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood glucose level at 120th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood TAS level at 120th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood TAS level at 120th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood TOS level at 120th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood TOS level at 120th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood glucose level at 180th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood glucose level at 180th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood TAS level at 180th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood TAS level at 180th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread and blood TOS level at 180th minute | One day
  Participants coming to the laboratory and eating control bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.
Whole wheat bread (added CMP and germ) and blood TOS level at 180th minute | One day
  Participants coming to the laboratory and eating test bread will have their capillary blood TOS measured with a calibrated glucometer at minute 0.

SECONDARY OUTCOMES:
Sociodemographic information form of participants eating whole wheat bread and whole wheat bread (added CMP and germ) | One day
  It is a form that questions information about the individual's health, education and economic status.
Determination of food consumption | One day
  Food consumption will be taken in order to evaluate differences between individuals that may affect the result. It covers a total of two days, one day before the 1st bread (standard whole wheat bread) and one day before the 2nd bread (test whole wheat bread), and the foods and beverages consumed by the individual are questioned.
Measurements of weight (kg) and height (cm) | 1 day
  Weight (kg) will be measured by Bioelectrical Impedance Analysis (BIA) body composition analyzer. Height (cm) will be measured using a stadiometer. The stadiometer comprises a rigid vertical backboard and a horizontal headboard running free, perpendicular to the backboard and without cross-play. The top of the head must be in contact with the headboard. After that, body mass index (BMI) will be calculated by using weight and height measurements. The formula is BMI = kg/m2 where kg is a person's weight in kilograms and m2 is their height in metres squared.
Measurements of Basal Metabolic Rate (kkal) | 1 day
  Basal Metabolic Rate (kkal) will be measured by Bioelectrical Impedance Analysis (BIA) body composition analyzer.
Measurements of Body Fat | 1 day
  Body Fat Mass (kg), Muscle Mass (kg), Visceral fat accumulation will be measured by Bioelectrical Impedance Analysis (BIA) body composition analyzer.
Measurements of Body Fluid | 1 day
  Total Body Fluid Mass (TBW) (L) (0.1 kg and 0.1%), Extracellular Fluid (ECW) (L) (0.1 kg), Intracellular Fluid (ICW) (L) (0.1 kg) will be measured by Bioelectrical Impedance Analysis (BIA) body composition analyzer. Edema wşll be calculated by the ratio of ECW/TBW.
Circumferences measurements | 1 day
  Waist and Hip Ratio can be measured and waist/hip ratio be calculated from participants eating both test and control bread.
Chemical analysis of test and control breads' protein content (%) | up to 8 weeks
  Chemical analysis were developed and the amount of both test and control bread containing 50 g carbohydrate and the amount of protein content (%) will be determined via analyses that will be carried at our university Food Chemistry Laboratory. Based on the results obtained, the amount of breads containing 50 g digestible carbohydrate will be calculated and produced.The Kjeldahl method will be applied to determine the total amount of nitrogen provided by the food. Protein content (%) is obtained by multiplying the total amount of nitrogen detected by the nitrogen factor determined according to the total organic nitrogen properties within the protein molecules. It is ensured that the test samples to be produced have more protein content than the standard.
Chemical analysis of test and control breads' moisture content (%) | up to 8 weeks
  Chemical analysis were developed and the amount of both test and control bread containing 50 g carbohydrate and the amount of moisture content (%) will be determined via analyses that will be carried at our university Food Chemistry Laboratory. Moisture content (%) will be based on the weight difference after drying in the oven at 105ºC until a constant weighing weight is reached. Moisture analysis in bread samples will be carried out after the bread is baked and cooled for 1 hour. The test samples to be produced are expected to contain moisture close to the standard.
Chemical analysis of test and control breads' specific volume (m3/kg or m3·kg-1) | up to 8 weeks
  Chemical analysis were developed and the amount of both test and control bread containing 50 g carbohydrate and the determination of specific volume (m3/kg or m3·kg-1) will be determined via analyses that will be carried at our university Food Chemistry Laboratory. The volumes of baked bread samples will be determined according to the rapeseed replacement method. The specific volume values of the bread samples produced are; It will be calculated by dividing the bread volume (cm3) to the bread weight (g). The test samples to be produced are expected to have a specific volume at least as much as that of control bread.
Chemical analysis of test and control breads' colorimetric assays (EBC) | up to 8 weeks
  Chemical analysis were developed and the amount of both test and control bread containing 50 g carbohydrate and the determination of colorimetric assays (EBC) will be determined via analyses that will be carried at our university Food Chemistry Laboratory.It will be carried out on the crust parts of the bread using the HunterLab brand hand-held color measuring device. L*, chroma (C), hue (h) values will be determined based on the CIE L*Ch* color system, which is one of the color definition models determined by the International Institute of Illumination (CIE). The test samples to be produced are expected to be close in color to control bread.
Chemical analysis of test and control breads' lipid content (%) | up to 8 weeks
  Chemical analysis were developed and the amount of both test and control bread containing 50 g carbohydrate and the amount of lipid content (%) will be determined via analyses that will be carried at our university Food Chemistry Laboratory. It will be carried out using the Soxhlet method. Approximately 4 g of bread samples will be weighed into a cellulose cartridge, covered with cotton and placed in the Soxhlet apparatus. At the end of the extraction using petroleum ether, the ether in the balloons will be evaporated and the oil content in the sample will be calculated. The test samples to be produced are expected to contain more unsaturated fatty acids than the control.
Chemical analysis of test and control breads' ash content (%) | up to 8 weeks
  Chemical analysis were developed and the amount of both test and control bread containing 50 g carbohydrate and the amount of ash content (%) will be determined via analyses that will be carried at our university Food Chemistry Laboratory. The samples will be weighed in a porcelain crucible that has previously been brought to a constant weight, and will be burned in a muffle furnace (Elektro-mag M1813, Turkey) at 550±5ºC until the residue becomes almost white in color. The % ash amount of the breads will be calculated by proportioning the sample mass remaining in the crucibles at the end of the burning process to the initial sample mass. The test samples to be produced are expected to contain more mineral substances than the control.
Chemical analysis of test and control breads' total phenolic content (mg GAE / g) | up to 8 weeks
  Chemical analysis were developed and the amount of both test and control bread containing 50 g carbohydrate and the amount of total phenolic content (mg GAE / g) will be determined via analyses that will be carried at our university Food Chemistry Laboratory. It will be determined by the Folin-Ciocalteau method. Sample extracts and Folin-Ciocalteau reagent prepared for this purpose will be used. 0.1 ml of extract will be mixed with 0.5 ml of Folin-Ciocalteu reagent (reagent: water mixture 1:10 v/v) and kept in the dark for 5 minutes. Then 0.4mL of saturated sodium carbonate solution and 4mL of pure water will be added. The mixture will be kept in the dark at room conditions for approximately 1 hour and the absorbance will be measured in a UV-VIS spectrophotometer at 760 nm. The result will be evaluated by calculating phenolic substance contents based on gallic acid equivalent. The test samples to be produced are expected to contain more polyphenols than the control.
Chemical analysis of test and control breads' antioxidant capacity (μg TE/g) | up to 8 weeks
  Chemical analysis were developed and the amount of both test and control bread containing 50 g carbohydrate and the amount of antioxidant capacity (μg TE/g) will be determined via analyses that will be carried at our university Food Chemistry Laboratory. 5 g sample will be taken from powdered defatted bread samples and mixed with 50 mL 80:20 methanol:water (v:v) for 30 minutes and then centrifuged at 4500 g for 15 minutes. 100 µL of the extracts will be taken into a cuvette and 3900 µL of DPPH (1,1-diphenyl-2-picrylhydrazyl radical) solution (2.36 mg/100 Mlmethanol) will be added and kept in the dark for 30 minutes. Absorbance measurements will be made on a spectrophotometer at 515 nm against the blank. Trolox calibration will be used to determine the activity value. The antioxidant value of the extracts will be stated as mMTrolox equivalent per kg. The test samples to be produced are expected to show more antioxidant properties than the control.
Chemical analysis of test and control breads' total starch analysis (g) | up to 8 weeks
  Chemical analysis were developed and the amount of both test and control bread containing 50 g carbohydrate and the amount of total starch analysis (g) will be determined via analyses that will be carried at our university Food Chemistry Laboratory. Total starch in the developed bread will be determined enzymatically according to the modified method of Goni et al. (1997). The test samples to be produced are expected to contain more starch than the control.
Chemical analysis of test and control breads' resistant starch (g) | up to 8 weeks
  Chemical analysis were developed and the amount of both test and control bread containing 50 g carbohydrate and the amount of resistant starch analysis (g) will be determined via analyses that will be carried at our university Food Chemistry Laboratory. Enzyme resistant starch will be determined in the samples using the "Megazyme resistant starch kit". For example, starch will be digested and converted into glucose with the help of α-amylase and amyloglucosidase enzymes. After adding ethyl alcohol to the samples, they will be centrifuged and the precipitated enzyme-resistant starch will be pelletized. After being dissolved with potassium hydroxide, the dissolved starch will turn into amyloglucose and glucose. Thus, the glucose formed will be determined spectrophotometrically. The test samples to be produced are expected to contain more resistant starch than the control.
Chemical analysis of test and control breads' in vitro starch digestion rate (%) and glycemic index | up to 8 weeks
  Starch digestion rate for breads will be expressed as the percentage of total starch hydrolyzed at incubation time intervals of 30 minutes, 60 minutes, 90 minutes and 120 minutes. The Hydrolysis Index (HI) will be derived from the ratio between the areas under the hydrolysis curve of the developed product and the reference sample (control wheat bread). From the obtained hydrolysis index, the estimated glycemic index (GI) will be calculated using the equation established by Goni et al. (1997). It is expected that the test samples to be produced will have a slower starch digestion rate and a lower glycemic index compared to the control.
Chemical analysis of test and control breads' moisture (baking) loss (%) | up to 8 weeks
  The moisture (baking) loss (%) value of bread samples will be based on the weight difference of the fixed dough weight (45 g) and the final product, baked bread samples. Baking loss (%) will be calculated with the formula = ((Dough weight-Bread weight)/Dough weight))*100. It is expected that the test samples to be produced will have a baking loss close to that of control bread.

CONTACTS AND LOCATIONS:
Overall Officials: Yüksel Özdemir, Prof., Principal Investigator — Head of Toros University Scientific Research Projects
Locations (1):
- Toros University, Mersin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tusat E, Parlak E, Yildirim G, Oztop K, Gulsen B, Ozdemir Y, Uysal Y. Impact of White Bread Fortified With Carob Molasses Pulp Flour and Wheat Germ on Glycemic Response and Antioxidant Capacity in Healthy Subjects. Food Sci Nutr. 2025 Dec 4;13(12):e71046. doi: 10.1002/fsn3.71046. eCollection 2025 Dec. PMID 41356220